CLINICAL TRIAL: NCT00329004
Title: A Phase I Dose Escalation Study of BMS-690514 in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Phase I Study of BMS-690514 in Patients With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA187-002
Record Dates: First submitted 2006-05-19; First posted 2006-05-24 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2009-08

CONDITIONS: Cancer; Tumor
Keywords: Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — BMS-690514

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: BMS-690514

INTERVENTIONS:
Drug: BMS-690514 — Tablets, Oral, up to 300 mg, once daily, up to 24 mos
  Other Names: panHER

SUMMARY:
The purpose of this research study is to determine the highest dose of the drug (BMS-690514) that can be safely given to patients with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 and older
* Diagnosis of any solid tumor
* ECOG performance status score 0-1
* Prior chemo-therapy, immunotherapy or radiotherapy with at least 4 weeks since the last treatment
* Treatment with VEGFR2 or HER1 TKI allowed but not both (for instance Avastin or Tarceva, but not both)

Exclusion Criteria:

* Treatment with other TKIs within the past 4 weeks
* Patients with brain metastasis
* Patients with centrally located squamous cell carcinoma of the lung
* Major gastrointestinal surgery which may affect absorption of the drug
* Any surgery within last 4 weeks
* History of thromboembolism
* Severe unmanageable diarrhea
* Subjects in Part B will have Non-Small Cell Lung Cancer (NSCLC)
* Part B/Cohort I erlotinib-naive subjects
* Part B/Cohort II subjects who have experienced disease progression while receiving erlotinib (erlotinib-resistant subjects)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2006-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Safety | results of weekly vital sign measurements, ECGs, laboratory tests and physical exams, echocardiograms every 8 weeks
Highest dose tolerated | continuous medical review of adverse event reports

SECONDARY OUTCOMES:
Effective dose or doses of BMS-690514 | tumor measurement by imaging every eight weeks. Continuous medical review of adverse event reports

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (2):
  - Indiana University Med Center, Indianapolis, Indiana
  - The University Of Texas Md Anderson Cancer Center, Houston, Texas
- Canada (2):
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario
- France (2):
  - Local Institution, Toulouse
  - Local Institution, Villejuif
- Local Institution, Barcelona, Spain

REFERENCES:
- [Derived] Soria JC, Baselga J, Hanna N, Laurie SA, Bahleda R, Felip E, Calvo E, Armand JP, Shepherd FA, Harbison CT, Berman D, Park JS, Zhang S, Vakkalagadda B, Kurland JF, Pathak AK, Herbst RS. Phase I-IIa study of BMS-690514, an EGFR, HER-2 and -4 and VEGFR-1 to -3 oral tyrosine kinase inhibitor, in patients with advanced or metastatic solid tumours. Eur J Cancer. 2013 May;49(8):1815-24. doi: 10.1016/j.ejca.2013.02.012. Epub 2013 Mar 13. PMID 23490650
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx